CLINICAL TRIAL: NCT05655377
Title: FitMi PD: an Affordable Home Therapy Device for Individuals With Parkinson's Disease
Brief Title: FitMi PD Home Therapy for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flint Rehabilitation Devices, LLC (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1R43AG071253-01 (NIH)
Record Dates: First submitted 2022-12-07; First posted 2022-12-19 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- At home exercise therapy with FitMi PD (Experimental): Participants will be instructed to use FitMi PD exercise system for three hours per week over 3-week period.
  Interventions: Device: FitMi PD

INTERVENTIONS:
Device: FitMi PD — Exercise using the motion sensing devices and a tablet computer

SUMMARY:
The investigators will run an at-home usability study of a newly developed home exercise device (FitMi PD) for individuals with Parkinson's disease. FitMi PD uses embedded sensors that can track and record the user's direction and degree of movement while performing exercises described on a computer.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate PD (Hoehn and Yahr stage I to III)
* Mini-Mental State Examination greater than 28

Exclusion Criteria:

* Age less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | At Home Exercise Therapy With FitMi PD
Started | 9
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | At Home Exercise Therapy With FitMi PD
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.11 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Successfully Used FitMi PD to Exercise at Home
Description: Number of participants who were successfully able to use the device at home to exercise over 3 week period.
Time Frame: Immediately Post-Treatment, an average of 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | At Home Exercise Therapy With FitMi PD
Number analyzed (Participants) | 9
Participants | 7

2. Secondary Outcome: Mini Mental State Examination (MMSE)
Description: A screening tool for assessing cognitive impairment. A maximum possible score of 30 is used to provide a picture of an individuals' present cognitive performance. A score of < 24 is the generally accepted cutoff indicating the presence of cognitive impairment.
  Levels of impairment have been classified as:
  None: score = 24-30 Mild: score = 18-24 Severe: score = 0-17
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | At Home Exercise Therapy With FitMi PD
Number analyzed (Participants) | 9
score on a scale | 30 (0.44)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | At Home Exercise Therapy With FitMi PD
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT05655377/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT05655377/ICF_001.pdf